CLINICAL TRIAL: NCT01201564
Title: Prospective Randomized Multicenter Trial Comparing Laparoscopic (IPOM) vs. Sublay Mesh Plasty for Umbilical Hernia in Adults
Brief Title: Comparative Study Matching Intraperitoneal Onlay Mesh (IPOM) and Sublay Mesh to Treat Umbilical Hernia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruiting problems
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPOM-46/10
Record Dates: First submitted 2010-07-19; First posted 2010-09-14 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Umbilical Hernia
Keywords: umbilical hernia,; wound complications,; mesh repair, IPOM,; quality of life,; sublay mesh repair,; recurrence rate
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraperitoneal onlay mesh repair (Active Comparator)
  Interventions: Procedure: intraperitoneal onlay mesh repair
- sublay mesh repair (Active Comparator)
  Interventions: Procedure: sublay mesh repair

INTERVENTIONS:
Procedure: intraperitoneal onlay mesh repair — The IPOM technique provides mesh positioning directly into the abdominal cavity onto the defect under laparoscopic control while in sublay position the mesh is placed directly behind des rectus muscle after small incision close to the belly button.
  Arms: intraperitoneal onlay mesh repair
Procedure: sublay mesh repair — The IPOM technique provides mesh positioning directly into the abdominal cavity onto the defect under laparoscopic control while in sublay position the mesh is placed directly behind des rectus muscle after small incision close to the belly button.
  Arms: sublay mesh repair

SUMMARY:
This study is designed to compare two techniques for operative care of umbilical hernia in adults regarding wound complications, wound side fluid collections, recurrence rate, postoperative pain, duration of hospitalization and quality of life. The IPOM technique provides mesh positioning directly into the abdominal cavity onto the defect under laparoscopic control while in sublay position the mesh is placed directly behind the rectus muscle after small incision close to the belly button.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patient age: ≥ 18 years
* elective surgery for umbilical hernia
* hernia diameter ≥ 1cm

Exclusion Criteria:

* previous history of median laparotomy
* navel site infection
* contraindication for general anaesthesia
* American Society of Anesthesiologists (ASA) score >IV
* pregnancy
* cirrhosis of the liver (CHILD B and C) and/or ascites
* cytostatic therapy
* incarcerated hernia
* recurrent hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2010-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
early wound complications | 30 days after operation
  * wound infection (with or without removal of the mesh)
  * wound necrosis
  * wound hematoma
late wound complications | 1 year after operation
  * wound infection (with or without removal of the mesh)
  * wound necrosis
  * wound hematoma

SECONDARY OUTCOMES:
complication rate perioperative | intraoperative complications will be recorded immediately after finishing the operation
  * major bleeding
  * bowel injury
duration of operation | the duration will be recorded immediately after finishing the operation
  measured in minutes according to operations protocol (duration cut - suture)
hospital stay | will be measured after discharge of the patient
  measured in days
umbilical hernia recurrence rate | 30 days
  the diagnosis of recurrence will be given by the surgeon clinically or due to ultrasound scan
umbilical hernia recurrence rate | 1 year
  the diagnosis of recurrence will be given by the surgeon clinically or due to ultrasound scan
umbilical hernia recurrence rate | 3 years
  the diagnosis of recurrence will be given by the surgeon clinically or due to ultrasound scan
umbilical hernia recurrence rate | 5 years
  the diagnosis of recurrence will be given by the surgeon clinically or due to ultrasound scan
navel site seroma | discharge day
  the diagnosis of seroma will be given by the surgeon clinically or by ultrasound scan and measured in ccm (height(cm) x width(cm)x length(cm))
navel site seroma | after 30 days
  the diagnosis of seroma will be given by the surgeon clinically or by ultrasound scan and measured in ccm (height(cm) x width(cm)x length(cm))
navel site seroma | after 1 year
  the diagnosis of seroma will be given by the surgeon clinically or by ultrasound scan and measured in ccm (height(cm) x width(cm)x length(cm))
complication rate postoperative | 30 day
  * trocar site hernia
  * enteral fistula
  * persistent pain
  * re-operation
complication rate postoperative | 1 year
  * trocar site hernia
  * enteral fistula
  * persistent pain
  * re-operation
complication rate postoperative | 3 years
  * trocar site hernia
  * enteral fistula
  * persistent pain
  * re-operation
complication rate postoperative | 5 years
  * trocar site hernia
  * enteral fistula
  * persistent pain
  * re-operation
pain score (Visual Analog Scale - VAS) | 24h post operative
  will be measured by the nurse according to Visual Analog Scale
pain score (Visual Analog Scale - VAS) | 48h post operative
  will be measured by the nurse according to Visual Analog Scale
pain score (Visual Analog Scale - VAS) | immediately before discharge
  will be measured by the nurse according to Visual Analog Scale
Quality of life (SF-36) | 1 day pre-operative
  patients will be asked to fulfill validated SF-36 questionnaire
Quality of life (SF-36) | 30 days postoperatively
  patients will be asked to fulfill validated SF-36 questionnaire
Quality of life (SF-36) | 1 year postoperatively
  patients will be asked to fulfill validated SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Oertli, Professor, Study Chair — Departement of General Surgery, University Hospital Basel, Switzerland; Oleg Heizmann, MD, Study Director — Departement of General,- Visceral- and Thoracic Surgery, Diakoniekrankenhaus Rotenburg (Wuemme), Germany; Daniel Matz, MD, Principal Investigator — Departement of General,- Visceral- and Thoracic Surgery, Diakoniekrankenhaus Rotenburg (Wuemme), Germany
Locations (3):
- Diakoniekrankenhaus Rotenburg (Wuemme) gGmbH, Rotenburg (Wümme), Lower Saxony, Germany
- Switzerland (2):
  - University Hospital Basel, Basel
  - Luzerner Kantonsspital, Lucerne

REFERENCES:
- [Background] Benhidjeb T, Benecke C, Strik MW. [Incisional hernia repair: sublay or intraperitoneal onlay mesh (IPOM)?]. Zentralbl Chir. 2008 Sep;133(5):458-63. doi: 10.1055/s-2008-1076954. Epub 2008 Oct 15. German. PMID 18924044
- [Background] Lau H, Patil NG. Umbilical hernia in adults. Surg Endosc. 2003 Dec;17(12):2016-20. doi: 10.1007/s00464-003-9027-7. Epub 2003 Oct 28. PMID 14574545
- [Background] Mayo WJ. VI. An Operation for the Radical Cure of Umbilical Hernia. Ann Surg. 1901 Aug;34(2):276-80. doi: 10.1097/00000658-190107000-00021. No abstract available. PMID 17861015
- [Background] Luijendijk RW, Hop WC, van den Tol MP, de Lange DC, Braaksma MM, IJzermans JN, Boelhouwer RU, de Vries BC, Salu MK, Wereldsma JC, Bruijninckx CM, Jeekel J. A comparison of suture repair with mesh repair for incisional hernia. N Engl J Med. 2000 Aug 10;343(6):392-8. doi: 10.1056/NEJM200008103430603. PMID 10933738
- [Background] Venclauskas L, Silanskaite J, Kiudelis M. Umbilical hernia: factors indicative of recurrence. Medicina (Kaunas). 2008;44(11):855-9. PMID 19124962
- [Background] Hilling DE, Koppert LB, Keijzer R, Stassen LP, Oei IH. Laparoscopic correction of umbilical hernias using a transabdominal preperitoneal approach: results of a pilot study. Surg Endosc. 2009 Aug;23(8):1740-4. doi: 10.1007/s00464-008-0177-5. Epub 2008 Nov 18. PMID 19015918
- [Background] Forbes SS, Eskicioglu C, McLeod RS, Okrainec A. Meta-analysis of randomized controlled trials comparing open and laparoscopic ventral and incisional hernia repair with mesh. Br J Surg. 2009 Aug;96(8):851-8. doi: 10.1002/bjs.6668. PMID 19591158
- [Background] Bullinger M. [Assessment of health related quality of life with the SF-36 Health Survey]. Rehabilitation (Stuttg). 1996 Aug;35(3):XVII-XXVII; quiz XXVII-XXIX. German. PMID 8975342